CLINICAL TRIAL: NCT03921359
Title: Effect of SMARTfit Training on Motor, Cognitive Functions and Brain Connectivity in Individuals With Parkinson's Disease: a Pilot Study
Brief Title: SMARTfit Training for Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: In compliance with research restrictions imposed due to the COVID-19 pandemic.
Sponsor: University of Southern California (Other)
Collaborators: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Charles Liu, Professor of Clinical Neurological Surgery, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HS-17-00928
Record Dates: First submitted 2019-01-08; First posted 2019-04-19 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Parkinson Disease; Exercise Training; Cognitive Change
Keywords: Parkinson Disease; Exercise Training; Cognitive function
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional physical training (Experimental): Participants assigned to this arm will receive the conventional physical training.
  Interventions: Behavioral: SMARTfit training; Behavioral: Conventional physical training
- SMARTfit training (Experimental): Participants assigned to this arm will receive the SMARTfit training.
  Interventions: Behavioral: SMARTfit training; Behavioral: Conventional physical training

INTERVENTIONS:
Behavioral: SMARTfit training — For SMARTfit training, participants receive three 1-hour training sessions per week for 8 weeks. During each week, participants will receive physical training focused on six tasks, which are the functional tasks individuals with PD commonly have difficulty with. The six tasks are paired into 3 pairs: (1) sit-to-stand and multi-plane locomotor tasks, (2) gait and reach & grasp, and (3) floor-to-stand; stand-to-floor and single limb standing. Participants will focus on practicing one pair of tasks during each session. There is an additional cognition component that can be manipulated using features provided by SMARTfit.
Behavioral: Conventional physical training — For conventional physical training, participants receive three 1-hour training sessions per week for 8 weeks. During each week, participants will receive physical training focused on six tasks, which are the functional tasks individuals with PD commonly have difficulty with. The six tasks are paired into 3 pairs: (1) sit-to-stand and multi-plane locomotor tasks, (2) gait and reach & grasp, and (3) floor-to-stand; stand-to-floor and single limb standing. Participants will focus on practicing one pair of tasks during each session.

SUMMARY:
This pilot study aims to investigate the effects of 8-week SMARTfit training versus conventional physical training on motor function, cognition and brain functional connectivity in individuals with PD. The investigators hypothesize that clinical and physical performance will improve after SMARTfit training more than after conventional physical training.

DETAILED DESCRIPTION:
Although Parkinson's disease (PD) has been mainly viewed as a movement disorder, the pathophysiology of declined motor function incorporates impairments of multiple systems, including sensory, motor and cognitive pathways. Specifically, it has been demonstrated that cognitive function may play an essential role in motor function for individuals with PD. Cognitive dysfunction involving set-shifting and attentional control has been found to be associated with movement slowness in performing a finger sequence task and freezing of gait. Furthermore, a recent rodent model indicates that cognitive dysfunction may occur prior to the onset of motor symptoms. Similarly human studies show that 25-30% individuals with PD exhibit cognitive impairments at the time of diagnosis. The overall evidence suggests that cognitive dysfunction may contribute to degraded motor function in PD. Interestingly, several studies demonstrate that aerobic exercise and resistance training can improve cognitive function in individuals with PD, indicating a tight interplay between motor and cognitive function. Targeting cognitive function by incorporating cognitive training into physical rehabilitation may be important for people with PD. Although there is mounting evidence for the benefits of physical exercise in PD, few studies investigate whether combining cognitive training with physical exercise can provide additional benefits than physical exercise alone. Thus, the purpose of this pilot study is to investigate the effect of SMARTfit training, a novel technology that provides an opportunity to combine physical training with cognitive training, in individuals with PD. The hypothesis is that SMARTfit training will promote greater motor and cognition improvements than conventional physical training. To test the above hypothesis, ten individuals with mild PD will receive both SMARTfit training and conventional physical training in a counterbalanced order with a washout period. For each training program, participants will receive a 1-hour training session 3 times per week for 8 weeks. The changes in disease biomarkers before and after training will also be explored.

ELIGIBILITY:
Inclusion Criteria:

1. 50-85 years of age
2. Diagnosis of idiopathic Parkinson's disease using the UK Brain Bank criteria (as determined by the study movement disorders neurologist) with Hoehn and Yahr stage 1-2
3. No contraindications to exercise including untreated cardiovascular disease or stroke
4. Medically stable and optimized on their medications
5. Able to ambulate independently with or without device
6. No other neurologic, neuromuscular, or orthopedic disease
7. No serious cognitive deficits and able to participate in the informed consent process
8. With medical clearance from primary care physician to participate in the physical therapy intervention
9. No contraindications for MRI

Exclusion Criteria:

1. Severe cardiac disease (New York Heart Association classification II-IV)
2. Systolic blood pressure reduction of greater than 20 mmHg with standing
3. A history of poorly controlled or brittle diabetes
4. A history of lower limb amputation
5. Been prescribed any new dopamine replacement medications or new mood stabilizer medications.
6. Presence of a lower limb non-healing ulcer
7. Montreal cognitive assessment score of less than 21
8. The presence of any medical condition which the investigator believes might present an unacceptable health risk to the subject should they participate in the study
9. Electrically, magnetically, or mechanically activated implant (such as cardiac pacemakers or intracerebral vascular clip)
10. Metal in any part of the body including metal injury to the eye
11. History of brain lesions (such as stroke), seizures, or unexplained spells of loss of consciousness
12. Pregnant or breast-feeding
13. With other neurologic, neuromuscular, or orthopedic disease that would interfere with ability to participate in exercise training
14. Currently participating in other studies

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-05-19 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Pre-post training change in Modified Physical Performance Test score (mPPT) | pre-assessment 1 (baseline), post-assessment 1 (8 weeks), pre-assessment 2 (after 2-month washout period after post-assessment 1, 16 weeks), post-assessment 2 (24 weeks)
  The mPPT is a 9-item test that assesses multiple dimensions of physical function (basic and complex activities of daily living) with different levels of difficulty. Participants will be asked to complete functional tasks (i.e. writing a sentence, simulated eating, lift a book and put it on a shelf, turning 360 degrees, 50-foot walking test, stair climbing etc.). Total score ranges from 0 to 36, with a higher score indicating better physical function.

SECONDARY OUTCOMES:
Pre-post training change in MDS-UPDRS score | pre-assessment 1 (baseline), post-assessment 1 (8 weeks), pre-assessment 2 (after 2-month washout period after post-assessment 1, 16 weeks), post-assessment 2 (24 weeks)
  The UPDRS is an assessment of Parkinson's disease severity and progress. The UPDRS has four sections. The first section assesses mental, mood, and behavioral changes. The second section assesses historical activities of daily living. The third section is the motor examination portion of the UPDRS and includes evaluations of tremor, rigidity, bradykinesia, gait, and postural instability. The fourth section evaluates complications of therapy including motor fluctuations and dyskinesias. Total score ranges from 0 to 260, with a higher score indicating greater disease severity.
Pre-post training change in Self-Efficacy for Exercise scale (SEES) | pre-assessment 1 (baseline), post-assessment 1 (8 weeks), pre-assessment 2 (after 2-month washout period after post-assessment 1, 16 weeks), post-assessment 2 (24 weeks)
  The SEE is to capture an individual's confidence in their ability to continue exercising in the face of barriers to exercise. The SEE consists of 9 items describing potential barriers to participation in exercise (e.g., "too busy with other activities," "did not enjoy exercise," "felt pain with exercise," "bored by the exercise"). For each item, participants circled a number from 0 ("not confident") to 10 ("very confident") that best described their belief that they could exercise 3 times a week for 20 minutes. Total score ranges from 0 to 90, with a higher score indicating higher self-efficacy for exercise.
Pre-post training change in trail-making test (TMT) | pre-assessment 1 (baseline), post-assessment 1 (8 weeks), pre-assessment 2 (after 2-month washout period after post-assessment 1, 16 weeks), post-assessment 2 (24 weeks)
  The Trail Making Test is a neuropsychological test of visual attention and task switching. It consists of two parts in which the participant is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. The test can provide information about visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning.
Pre-post training change in Parkinson's Disease-Cognitive Rating Scale (PDCRS) | pre-assessment 1 (baseline), post-assessment 1 (8 weeks), pre-assessment 2 (after 2-month washout period after post-assessment 1, 16 weeks), post-assessment 2 (24 weeks)
  The PDCRS is is a valid, reliable and useful neuropsychological battery designed to cover the full spectrum of cognitive defects associated with PD. The PDCRS includes 10 'subcortical-type' items (attention, working memory, Stroop test, four verbal fluencies, immediate and delayed verbal memory, clock drawing), and two 'cortical-type' items (naming, copy of a clock). Total score ranges from 0 to 204, subcortical score from 0 to 174, and cortical score from 0 to 30, with higher scores indicating a better functioning.
Pre-post training change in Quotient system test | pre-assessment 1 (baseline), post-assessment 1 (8 weeks), pre-assessment 2 (after 2-month washout period after post-assessment 1, 16 weeks), post-assessment 2 (24 weeks)
  The Quotient test is an innovative device that objectively measures three domains of cognition: hyperactivity, inattention and impulsivity.
Pre-post training change in functional connectivity | pre-assessment 1 (baseline), post-assessment 1 (8 weeks), pre-assessment 2 (after 2-month washout period after post-assessment 1, 16 weeks), post-assessment 2 (24 weeks)
  Participants will receive resting state fMRI, in which they will be instructed to keep their eyes open fixation on a projected image of a white cross on a black background. Participants will also receive task-based fMRI, in which they will be asked to perform a word-color Stroop task.
Pre-post training change in EEG delta (2.5-4 Hz) bandpower | pre-assessment 1 (baseline), post-assessment 1 (8 weeks), pre-assessment 2 (after 2-month washout period after post-assessment 1, 16 weeks), post-assessment 2 (24 weeks)
  A 19-channel EEG acquisition system will be used in recording. Participants will be instructed to sit quietly with eyes closed whilst wearing a skull cap.
Change in the concentration of α-synuclein and DJ-1 | pre-assessment 1 (baseline), post-assessment 1 (8 weeks), pre-assessment 2 (after 2-month washout period after post-assessment 1, 16 weeks), post-assessment 2 (24 weeks)
  A venous blood sample of up to 40 ml will be obtained from participants.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Liu, MD, PhD, Principal Investigator — University of Southern California
Locations (1):
- USC Center for Neurorestoration, Los Angeles, California, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/59/NCT03921359/Prot_SAP_000.pdf